CLINICAL TRIAL: NCT01827085
Title: Time to Intubation in Obese Patients. A Comparison Between Macintosh Laryngoscope and Stortz Video Laryngoscope
Brief Title: Time to Intubation (TTI) of Obese Patients. A Comparison Macintosh Laryngoscope and Stortz Video Laryngoscope
Acronym: TTI
Status: Completed | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Alex de Leon, PhD, Örebro University, Sweden
Other Study IDs: EPN2012/015
Record Dates: First submitted 2013-03-26; First posted 2013-04-09 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Macintosh laryngoscope: Patients will be intubated with a conventional Machintosh laryngoscope
  Interventions: Device: Conventional Macintosh laryngoscope
- Videolaryngoscope: Intubation with Stortz video laryngoscope
  Interventions: Device: Stortz videolaryngoscope

INTERVENTIONS:
Device: Conventional Macintosh laryngoscope
  Groups: Macintosh laryngoscope
Device: Stortz videolaryngoscope
  Groups: Videolaryngoscope

SUMMARY:
The purpose of the study is to investigate wether the use of the Stortz video laryngoscope will render in shorter time for the intubation of obese patients compared with the use of a conventional Macintosh laryngoscope.

DETAILED DESCRIPTION:
Obese patients are prone to develop desaturation soon after initiation of anaesthesia compared to patients of normal body weight. It is therefore important to keep the time from when spontaneous breathing to when the airway is secured with a orotracheal tube as short as possible. We will therefore investigate if it is possible to shorten this time by using a Stortz videolaryngoscope.

Patients 18-60 years with ASA grade 1-3 and BMI < 35 that turn up for planned surgery that demands the use of orotracheal tubing and controlled ventilation will be randomly and consecutively enrolled in either of two groups. Patients in both groups will be anaesthetised with the same combination of drugs using Propofol and Remifentanyl or Fentanyl for induction of sleep, combined with Rocuronium for muscle relaxation.

After the induction and relaxation the intubation will be facilitated using either of two laryngoscopes. In the first group a conventional Macintosh laryngoscope, and in the second group a Stortz videolaryngoscope will be used. The time to intubation is defined as the time from grabbing the laryngoscope to when the tube has been inserted and end-tidal carbon dioxide appears on the monitor. Our hypothesis is that we will be able to achieve a faster intubation with the use of videolaryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Obesity defined as BMI > 35
* ASA 1-3

Exclusion Criteria:

-known or suspected difficult airway

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In-patients from the University hospital of Orebro who will go through planned surgery
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Time to intubation seconds (s) | Up to 1 minute

SECONDARY OUTCOMES:
Presence and level of postoperational throat pain | 1 hour to 96 hours postoperative
  If throat pain is present, we will use a visual analogue scale to evaluate the level of throat pain 1h, 24h, 72h and 96h after extubation.
Ease of intubation | Two minutes
Incidence of trauma in each group | Two minutes
Number of attempts of intubation | Two minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaethesia and Intensive Care, University Hospital Örebro, Örebro, Sweden